CLINICAL TRIAL: NCT00713180
Title: Determinants of Pterygium Occurrence and Recurrence in a Rural African Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anguria, Peter, M.D. (Individual)
Responsible Party: Anguria Peter, Mankweng Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Research laboratory
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2008-08

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Pterygium free participants
- 2 (Experimental): Pterygium participants
  Interventions: Procedure: Pterygium excision followed by grafting

INTERVENTIONS:
Procedure: Pterygium excision followed by grafting — Pterygium will be excised followed by either free conjunctival or limbal conjunctival graft obtained from the upper part of the globe. The graft will be kept in place by sutures
  Arms: 2

SUMMARY:
The aim of the study is to find out why pterygium occurs and recurs in a rural African population. Participants will be interviewed on personal and lifestyle information, family history of pterygium, environmental exposure and history of previous eye inflammation. They will undergo eye examination and photography. Those with pterygium will be operated on to remove pterygium and followed up to detect any recurrence and complications of surgery. The excised pterygium will be examined pathologically and genetically; participant's blood will also be examined genetically. Data will be analyzed for statistically significant differences in findings between pterygium and pterygium free participants.

The study hypothesis is that multiple factors are responsible for the occurrence and recurrence of pterygium in a rural african population.

ELIGIBILITY:
Inclusion Criteria:

1. Pterygium at least 1.5mm in extent
2. Both male and female
3. Age range 21-65 years
4. Consenting to participate in study
5. Unilateral and bilateral pterygium
6. All grades of pterygium

Exclusion Criteria:

1. Previous cataract, corneoscleral and glaucoma surgery or corneoscleral trauma and corneolimbal scars
2. Pseudopterygium or signs of malignancy on pterygium
3. Recurrent pterygium
4. Sufferers of collagen vascular disease, scleritis or diabetes -

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 355 (Estimated)
Dates: Start 2008-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
None recurrence of pterygium | 6 months of follow up after operation

SECONDARY OUTCOMES:
corneal scarring | 6 months of follow up
tenon's granuloma | 6 months of follow up
graft retraction | one month of follow up
Graft haematoma | one week of follow up
Graft hyperaemia | 3 months of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Peter Anguria, MMed, Principal Investigator — Mankweng Hospital
Locations (1):
- Mankweng Hospital, Polokwane, Limpopo, South Africa